CLINICAL TRIAL: NCT06211933
Title: Phase I/II Study Evaluating the Safety and Efficacy of the HIFU Technique in Patients With Unresectable Pancreatic Tumor
Brief Title: Evaluation of the High Intensity Focused Ultrasound (HIFU) Technique for Patients With Unresectable Pancreatic Tumor Treatment (PULS)
Acronym: PULS
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Following a decision by the industrial partner, it was decided to permanently close the study to new participants.
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET23-247 (PULS)
Record Dates: First submitted 2023-12-20; First posted 2024-01-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-Resectable Pancreas Carcinoma
Keywords: Oncology; Phase I; Phase II; Phase I/II; HIFU; High Intensity Focalised Ultrasounds; Efficacy; Safety; Medical Device
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: HIFU intervention at day 0 for each patient included.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFU intervention (Experimental): HIFU intervention
  Interventions: Procedure: HIFU intervention

INTERVENTIONS:
Procedure: HIFU intervention — HIFU intervention on non resectable pancreatic lesions at day 0 for each patient included

SUMMARY:
This is a phase I/II, multicenter trial for patients with locally advanced and unresectable pancreatic tumours :

* A Phase I evaluating the tolerance of intraoperative High Intensity Focused Ultrasound (HIFU) intervention on the pancreatic lesion.
* A non-randomized Phase II evaluating the preliminary efficacy of the HIFU intervention on the pancreatic lesion.

Patients included in Phase I will be monitored and included in the Phase II evaluation.

DETAILED DESCRIPTION:
The PULS study is designed for patients with a locally advanced tumour of the pancreas (known as pancreatic adenocarcinoma) that has previously been treated with several cycles of chemotherapy and cannot be removed by surgery.

Pancreatic adenocarcinomas are often diagnosed at an advanced stage and only 15% to 20% of patients are candidates for surgery to remove the tumour. In the remaining cases, around a third of patients have metastatic disease at the time of diagnosis. The remaining third have locally advanced pancreatic cancer. In these cases, chemotherapy with or without radiotherapy is the standard treatment. The low proportion of patients who can benefit from surgery and the poor response to chemotherapy make the development of new treatments vital and urgent.

For locally advanced cancers, we want to develop and evaluate a new form of treatment based on a medical device using high intensity focused ultrasound (HIFU), after chemotherapy.

HIFU is a recent technology that uses therapeutic ultrasound. All HIFU procedures currently performed are carried out using an extracorporeal approach.

The aim of this research is therefore to assess the safety and efficacy of HIFU ablation of locally advanced pancreatic tumours.

This trial is a two stages (phase I and II) open label non comparative study. The first step of this study is to evaluate the safety of the HIFU intervention on 3 to 6 patients included. Patients will be included one by one, with a safety committee after each intervention. The total number of patients included in phase I will depend on the complications rate : If no serious complications are observed among the first 3 patients treated, the phase II study can begin. If a serious complication is observed, 3 additional patients will be included in phase I. The transition to phase II will be effective if a maximum of 1 complication out of the 6 patients included is observed. In the other cases, if at least 2 serious complications are observed for 3 to 6 patients included, the study will be definitively stopped.

The second step of this study is to evaluate the efficacy of the HIFU intervention on 26 patients including the patients of phase I.

Each patient will be follow for two years after the HIFU intervention. Un update of vital status will be made annually until the last patient's last visit.

Sample size was thus evaluated by analogy with an A'Hern's. If at least 14 successes are observed among 26 patients, HIFU treatment will be considered of interest.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the day of consenting to the study
* Patient with histologically confirmed locally advanced (unresectable) pancreatic adenocarcinoma according to the National Comprehensive Cancer Network (NCCN) 2020 classification
* Unifocal pancreatic lesion with a maximum diameter of 4 cm
* Non-progressive disease after 4 months of first-line chemotherapy or after 2 months of chemotherapy in case of limiting toxicity contraindicating continuation of chemotherapy;
* Preoperative imaging including CT-scan, MRI of the liver and Positron Emission Computed Tomography scan (PET-CT scan) (except for absolute medical contraindications), within 4 weeks prior to HIFU treatment
* Eastern Cooperative Oncology Group performance status ≤ 2
* Adequate hematologic parameters defined by platelets ≥ 100 Giga/l and hemoglobin ≥ 8 g/dl
* Ability to understand and willingness for follow-up visits
* Patient affiliated to a health insurance scheme (or beneficiary of such a scheme)
* Signed and dated informed consent document indicating that the patient has been informed of all aspects of the trial prior to enrolment

Exclusion Criteria:

* Local recurrence of previously operated pancreatic cancer
* Metastatic pancreatic carcinoma
* History of major pancreatic resection
* Chemotherapy completed less than 2 weeks ago
* History of radiotherapy to the pancreas
* Pregnant women
* Possibility of R0 resection with venous reconstruction
* Inability to undergo study follow-up for geographical, social or psychological reasons
* Patient requiring tutorship or curatorship or patient deprived of liberty
* Patient under psychiatric care against his wishes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Tolerance profile of HIFU intervention | Up to 30 days after HIFU intervention
  The tolerance of HIFU intervention will be assessed by the number of patients presenting at least one serious complication during the first 30 days after HIFU intervention. A serious complication corresponds either to any grade 3 or more complication according Clavien-Dindo classification or any vascular complication treated by interventional radiology
Survival rate at 12 months after HIFU intervention | Up to 12 months after HIFU intervention
  The efficacy of treatment will be assessed by the proportion of patients alive 12 months after HIFU treatment

SECONDARY OUTCOMES:
Tumor ablation rate by HIFU | Up to 28 days after inclusion
  The tumor ablation rate by HIFU is defined by the volume of the area destroyed by HIFU compared to the volume of the pancreatic cancer on the imaging
Intra-operative and post-operative complications linked to the HIFU intervention | Up to 3 months after HIFU intervention
  The Intra-operative and post-operative complications linked to the HIFU intervention will be evaluated by the number of patients with at least one complication according to Clavien Dindo classification appeared during HIFU intervention and until 3 months after HIFU intervention
Feasibility of HIFU intervention | Up to 28 days after inclusion
  The feasibility of HIFU intervention will be evaluated by the rate of patients who were able to benefit from HIFU intervention. The reasons for non-completion will be described.
Progression-Free Survival (PFS) | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first or until the date of the last update for patients without progression, assessed up to 60 months after inclusion
  The Progression-Free Survival (PFS) will be defined as the time from the date of HIFU intervention to the date of first documented disease progression or the date of death due to any cause or until the date of the last update for patients without progression
Local Progression-Free Survival (local PFS) | From date of inclusion to the date of first disease progression or death or last update, assessed up to 60 months
  The local Progression-Free Survival (local PFS) will be defined as the time from the date of HIFU intervention to the date of first local progression
Overall Survival (OS) | From date of inclusion to the date of death or date of last update, assessed up to 60 months
  The Overall Survival (OS) will be defined as the time from date of HIFU intervention to the date of death, from any cause. Patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Length of hospitalization | From date of HIFU intervention to the date of discharge from hospitalization, assessed up to 3 months
  The length of hospitalization will be calculated by number of days from the date of the HIFU intervention until the date of discharge from hospitalization
Rehospitalization rate during the first 30 days after HIFU intervention. | From the date of HIFU intervention to 30 days after HIFU intervention
  The rehospitalization rate during the first 30 days after HIFU intervention will be calculated by the number of patients rehospitalized during the first 30 days after HIFU intervention compared to the total number of patients who received HIFU intervention
Rate of secondary resectability | From date of HIFU intervention to the date of last patient's last visit, assessed up to 60 months
  The secondary resectability will be calculated by the number of patients eligible for curative pancreatic resection following HIFU intervention compared to the total number of patients who received HIFU intervention
Incidence and severity of adverse events | From the date of intervention to the date of last patient's last visit, assessed up to 60 months.
  Descriptive statistics will be used to describe the tolerance profile to HIFU intervention. The incidence and severity of adverse events (AEs), HIFU procedure-related AEs, Serious Adverse Events (SAEs), and deaths will be graded according to the latest version of the Common Terminology Criteria for Adverse Events (CTCAE) classification.
Quality of Life (QoL) | From the date of inclusion to 6 months after HIFU intervention
  The patient's Quality of Life (QoL) will be assessed using the European Organisation for Research and Treatment of Cancer (EORTC) Quality Of Life Questionnaire C30 file. The questionnaire includes 30 questions whose scores will be calculated at each time point according to the scoring manuals of EORTC. Descriptive statistics will be used to evaluate baseline scores and evolution of scores from inclusion to each time point. The QoL data will also be presented graphically.
  Questions 1 to 28 will be evaluated by a score from 1 to 4, 1 being the best outcome and 4 the worse and questions 29 and 30 will be evaluated by a score from 1 to 7, 1 being the worse outcome and 7 being the best.
Clinical benefice rate regarding pain | From the date of inclusion to the date of last patient's last visit, assessed up to 60 months.
  The clinical benefice rate regarding pain will be calculated by the number of patients showing an improvement in pain from inclusion to the end of study, compared to the total number of patients who received HIFU intervention. Pain will be assessed by an analog visual scale (0 to 10 scale, 0 being the best score and 10 the worse).
Clinical benefice rate regarding weight | From the date of inclusion to the date of last patient's last visit, assessed up to 60 months.
  The clinical benefice rate regarding weight will be calculated by the number of patients showing an improvement in weight (in kilograms) from inclusion to the end of study, compared to the total number of patients who received HIFU intervention. A 10% or more increase of weight will be considered as a weight improvement.
Clinical benefice rate regarding performance status | From the date of inclusion to the date of last patient's last visit, assessed up to 60 months.
  The clinical benefice rate regarding performance status will be calculated by the number of patients showing an improvement in performance status from inclusion to the end of study, compared to the total number of patients who received HIFU intervention. Performance status will be assessed by the Eastern Cooperative Group of Oncology (ECOG) score.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Estaing, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes